CLINICAL TRIAL: NCT06537778
Title: Perioperative Use of Atosiban for Ultrasound-indicated Cerclage to Reduce Spontaneous Preterm Birth(sPTB)
Acronym: sPTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Li Qin, Principal Investigator, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-043; NCT06399965 (obsolete NCT alias)
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cerclage; Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — atosiban; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- atosiban (Experimental)
  Interventions: Drug: Atosiban
- normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Atosiban — Women in the atosiban group received i.v. atosiban (Manufacturer: Pfizer, Germany) 30 min before the surgery with a bolus dose of 6.75 mg, and the infusion was continued with an infusion rate of 18 mg/h for 3 h. The dose of atosiban was then reduced to 6 mg/h for another 45 h.
  Arms: atosiban
Drug: Normal saline — Participants in the placebo group received only normal saline infusion for the same duration as atosiban group.
  Arms: normal saline

SUMMARY:
After ultrasound-indicated cerclage, some pregnant women still experience sPTB, and there is controversy regarding the use of tocolytic agents during the perioperative period to reduce the incidence of sPTB. In this study, the investigators employed a randomized double-blind method to investigate whether the use of atosiban during the perioperative period can reduce the incidence of sPTB before 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

* (i) Viable singleton gestation between 14 0/7 and 23 6/7 weeks of gestation.
* (ii) Previous history of miscarriage or preterm labor in mid-pregnancy.
* (iii) Transvaginal ultrasound examination showed that the cervix is 25mm or less at gestations less than 24 weeks.

Exclusion Criteria:

* (i) Women with uterine contractions.
* (ii) Vaginal bleeding.
* (iii) Symptoms of chorioamnionitis.
* (iv) Medically indicated PTB (severe preeclampsia, placental abruption, preterm premature rupture of membranes).
* (v) Major structural or chromosomal abnormalities.
* (vi) Contraindication to atosiban.
* (vii) Had received atosiban or any tocolytic agents within 7 days before their presentation.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Rate of sPTB | up to 34 weeks
  Rate of sPTB before 34 weeks of gestation

SECONDARY OUTCOMES:
Rate of preterm delivery <28 or <32 weeks gestation | up to 32 weeks
  Rate of preterm delivery <28 or <32 weeks gestation
Gestational latency after cerclage placement (days) | through study completion, an average of 1 year
  Gestational latency after cerclage placement (days)
Rate of preterm premature rupture of membranes | through study completion, an average of 1 year
  Rate of preterm premature rupture of membranes
Gestational age at delivery (weeks) | through study completion, an average of 1 year
  Delivery weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Women and Children's Hospital of Chongqing Medical University, Chongqing, Chognqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No
Based on the requirements of the ethics committee, the data from this study cannot be shared.